CLINICAL TRIAL: NCT04128189
Title: Safety and Immunogenicity of Shingrix in Renal Transplant Recipients
Brief Title: Shingrix in Renal Transplant Recipients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-0005
Record Dates: First submitted 2019-09-25; First posted 2019-10-16 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant Recipient Response to Shingrix Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transplanted subject (Active Comparator): In addition to receiving standard dose (2) of Shingrix prior to transplantation, participant may receive a 3rd dose several months after transplantation if they meet criteria related to no rejection.
  Interventions: Biological: Shingrix
- Non-Transplanted subject (Sham Comparator): Receives standard Shingrix dose (2), but not transplanted within 16 month time frame post-dose, so does not receive additional Shingrix dose.
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: Shingrix — Both arms receive standard 2 doses of Shingrix. Transplanted subjects may receive 3rd dose.

SUMMARY:
This study evaluates the safety and immune response of the Shingrix vaccine in kidney transplant recipients. Participants on the waiting list for kidney transplant will be given the standard 2 doses of Shingrix. Those participants who have been transplanted by 16 months, may be given a 3rd dose of Shingrix.

DETAILED DESCRIPTION:
Herpes Zoster (HZ) is a common complication of kidney transplant because of the immune suppressive drugs necessary to prepare the recipient for the transplanted organ and to protect it from rejection. The use of the live vaccine, Zostavax, in transplant recipients is contraindicated due to their impaired immune status. This study is being done to determine vaccine responses to the FDA approved shingles vaccine, Shingrix, in patients with chronic renal failure eligible for kidney transplant. Persistence of immune responses after kidney transplantation, and immunologic advantage of a third dose of Shingrix to renal transplant recipients will be assessed. Additionally, safety, tolerability, and occurrence of HZ will be evaluated. 60 participants will be enrolled from the renal transplant services at University of Colorado Anschutz Medical Campus.

ELIGIBILITY:
Inclusion Criteria:

* On the waiting list at the participating institutions for renal transplantation with anticipated transplantation to occur at > 3 months to 16 months after listing.
* Female subjects of non-childbearing potential (tubal ligation, hysterectomy,ovariectomy or post-menopausal
* Female subjects of childbearing potential who have practiced adequate contraception for 30 days prior to vaccination, have a negative pregnancy test on day of vaccination, and have agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccine series

Exclusion Criteria:

* Therapy in the pre-transplant period that in the opinion of the investigator is immune suppressive
* Herpes Zoster in prior 3 years
* Herpes zoster vaccine or varicella vaccine within 3 years of study entry
* Any positive cPRA score prior to enrollment
* Acute illness at the time of vaccination which in the opinion of the investigator will alter immune response
* Any other active immunosuppressive or immunodeficient condition resulting from disease (e.g. malignancy, HIV, or a medical therapy).
* Allergy to any of the components of Shingrix
* No investigational drugs from 30 days before enrollment or planned during the study.
* No non-live vaccines within the 2 weeks prior to any dose of Shingrix or until 30 days after any dose of Shingrix. No live virus vaccines within 4 weeks prior to any dose of Shingrix or until 30 days after any dose
* Pregnant or lactating female
* Multi-organ transplantation
* Travel time from study site that is more than 2 hours for visit or transport of fresh blood samples

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Immunology - Glycoprotein E(gE)-specific antibody and cell mediated immunity (CMI) will be measured. | 12 months after vaccination
  The kinetics and magnitude of antibody and CMI responses will be compared to immunologic data previously determined during studies of immune competent subjects.
Safety information acquisition - Adverse events (AEs) | Adverse event data collected for 30 days after each vaccine dose.
  Safety and tolerability data about local and systemic adverse events will be collected via vaccine diaries.
Ascertaining occurrence of HZ in vaccinees | At every contact from enrollment up to Month 36
  Subjects will be asked to notify study team and to complete an HZ questionnaire should they develop herpes zoster during the study.
Safety information acquisition - Serious Adverse Events (SAEs) and potential immune-mediated diseases (pIMDs) | SAEs and pIMD data collected from enrollment up to 12 months after Visit 4
  Subjects will be queried about SAEs and pIMDs at every contact.

SECONDARY OUTCOMES:
Immunologic vaccine responses in patients with chronic renal failure | 1 month after 2nd dose of Shingrix.
  gE-Specific IL2 SFC/10; interleukin-2 = IL2, spot forming cells = SFC

CONTACTS AND LOCATIONS:
Overall Officials: Myron J Levin, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No